CLINICAL TRIAL: NCT05684393
Title: Anatomy-based Fitting in Unexperienced Cochlear Implant Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dominik Riss (Other)
Responsible Party: Sponsor-Investigator, Dominik Riss, Assoc.-Prof. Priv.-Doz. Dr. med., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2131/2021
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Influence of Anatomy Based Frequency Mapping on Speech Outcomes and Hearing Related Measures

STUDY DESIGN:
Intervention Model Description: The performance with the CI is investigated over time in two groups of freshly implanted CI users. The first group is fitted using the standard frequency-band distribution as implemented in MAESTRO 9 fitting software. In the second group of users, an anatomy-based frequency distribution is used as per anatomy-based fitting in MAESTRO 9.
Who Masked: Participant, Investigator
Masking Description: double blinded design: both the participant and the investigator have no information about the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anatomy based fitting (Experimental)
  Interventions: Other: frequency distribution type
- Standard fitting (Active Comparator)
  Interventions: Other: frequency distribution type

INTERVENTIONS:
Other: frequency distribution type — One group is fitted using channel filterbank frequency distribution based on anatomy data extracted from post-OP CT measurements. The second (control) group is fitted with the standard frequency distribution used in MAESTRO 9 fitting software.

SUMMARY:
The present study investigates CI users' potential differences in speech tests, other performance measures (i.e. pitch-matching, perception of timbre and melodic intervals, consonance perception), and patient-reported outcome (i.e. questionnaires) between the clinical fitting map and anatomy-based fitting in two groups of CI users (one with standard fitting and one with anatomy-based fitting).

ELIGIBILITY:
Inclusion Criteria:

* Post-lingual onset of severe to profound sensory-neural hearing loss in the implanted ear(s)
* Post-OP CT scan of the CI electrode available
* Subject implanted with MED-EL cochlear implant(s)
* Subjects received a Flex28, FlexSoft and Standard electrode
* Subject planned to receive a SONNET 2 or RONDO 3 audio processor on the newly implanted side
* Audio processor not yet activated on the newly implanted side
* The most apical active electrode contact has to be inserted at least 450°
* Minimum of 10 active channels can be activated
* Fluent in the language of the test centre
* Signed and dated ICF before the start of any study-specific procedure

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* EAS user (user of an EAS audio processor)
* Implanted with C40+, C40X and C40C
* Implanted with an ABI or Split electrode array
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Word recognition score (WRS) | 6 months
  Percentage of correctly understood monosyllabic words from a list.

SECONDARY OUTCOMES:
Speech reception threshold (SRT) | 6 months
  German matrix sentence test - speech to noise ratio in dB.
Pitch ranking | 6 months
  Difference of the mean ranks for a set of frequencies presented to the tested CI ear and the reference ear.
Perception of timbre | 6 months
  Visual Analog Scale ratings describing the difference in timbre between the tested CI ear and the reference ear when listening to audio.
Phoneme categorization | 6 months
  Shape of the psychometric function describing the perception of the /s/-/ʃ/ continuum.
Consonance/difference rating | 6 months
  The degree of modulation of the pleasantness-score across the individual intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria